CLINICAL TRIAL: NCT00714454
Title: 5% Sodium L-Ascorbyl-2-Phosphate Lotion for the Treatment of Acne Vulgaris: A Double-Blind, Placebo Controlled Trial
Brief Title: 5% Sodium L-Ascorbyl-2-Phosphate Lotion for the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Ikeno Clinic (Unknown)
Other Study IDs: 97269358-APS
Record Dates: First submitted 2008-07-03; First posted 2008-07-14 (Estimated); Last update posted 2008-07-14 (Estimated); Status verified 2008-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APS (Active Comparator)
  Interventions: Other: APS Topical Lotion
- Vehicle (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: APS Topical Lotion
  Arms: APS
Other: Placebo
  Arms: Vehicle

SUMMARY:
12-week study to compare the efficacy and safety of a course of a twice daily treatment with APS in the form of a lotion to its vehicle for the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Subject has read, understood, and signed appropriate informed consent, photo consent, and HIPAA consent in their own language.
* Subject has visible mild to severe acne, as assessed by the investigator.
* Subject will be available and willing to return for follow-up visits.
* Subject agrees not to use any other acne treatment products during the study.
* Subject is otherwise healthy, non-febrile, and is not suffering from an infection likely to require antibiotic therapy during the study period.
* Subject or guardian must be able to understand the new HIPAA regulations and sign the HIPAA form.
* Subject is between the ages of 18 and 39.
* Subject agrees and understands that APS or its vehicle is to be applied to the subject twice daily for 12 weeks; no other topical or systemic medication affecting the course of acne and/or evaluability is to be used during the study.
* Subject agrees to use only the cleanser, moisturizer with sunscreen, and treatment provided by the study site for the duration of the study.
* Subject understands and agrees that he/she can not be treated with a systemic antibiotic for acne during the study.
* Subject agrees he/she will not use an acne topical treatment for two weeks prior to Day 0.

Exclusion Criteria:

* Subject or guardian has not signed informed consent, photo consent or HIPAA form.
* Subject is suffering from a condition likely to require medical attention, including administration of oral or systemic antibiotics, oral or systemic corticosteroids, or any other treatment which in the opinion of the investigator could influence the results of the study.
* Subject is pregnant or lactating.
* Subject is suffering from an abnormal skin condition not usually associated with acne.
* Subject will not be available for follow-up visits.
* Subject has been previously enrolled in any clinical study in which treatment was received within the past 30 days.
* Subjects without comedones, papules, pustules, or nodules.
* Subject has a history of hypersensitivity to any other ingredients of the study lotion.
* Subject has a history of anaphylaxis.
* Subject is not able to avoid excessive sun exposure.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Heather Woolery-Lloyd, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Cosmetic Center, Miami Beach, Florida, United States